CLINICAL TRIAL: NCT06863350
Title: Efficacy and Safety of Percutaneous Foramen Ovale Closure in Adult Patients with Drug-resistant Epilepsy and Patent Foramen Ovale: a Randomized Controlled Trial
Brief Title: Percutaneous Repair for Drug - Resistant Epilepsy by Intervention of Closing the Patent Foramen Ovale（PREDICT-PFO Trial）
Acronym: PREDICT-PFO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Bo Zhang, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX20242572; ZYYC23011 (Other Grant/Funding Number: Lei Chen)
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy (treatment Refractory)
Keywords: patent foramen ovale; epielpsy
MeSH Terms: conditions — Epilepsy; Foramen Ovale, Patent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operation group (Experimental): patent foramen ovale closure
  Interventions: Device: patent foramen ovale closure
- control group (No Intervention)

INTERVENTIONS:
Device: patent foramen ovale closure — patent foramen ovale closure
  Arms: Operation group

SUMMARY:
Patent foramen ovale (PFO) is the most common cause of right-to-left shunt (RLS) in the adult heart, with a prevalence of approximately 25% in the general population. Extensive research has demonstrated an association between PFO and neurological conditions such as cryptogenic stroke, migraine, and sleep apnea syndrome, and it is even considered a potential root cause of these disorders. However, the mechanisms by which PFO contributes to neurological diseases remain unclear. In our preliminary clinical work, we have observed a strong correlation between PFO and epilepsy, and PFO closure has shown some efficacy in reducing seizure frequency. The aim of this study is to further investigate the efficacy and safety of PFO closure in patients with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years, with no gender restrictions;
2. Diagnosis of epilepsy in accordance with the International League Against Epilepsy (ILAE) criteria (2014 edition);
3. Drug-resistant epilepsy, defined as failure to achieve sustained seizure freedom despite appropriate selection and tolerability of at least two antiseizure medications (monotherapy or combination therapy) for a minimum of six months;
4. Diagnosis of patent foramen ovale (PFO) meeting the criteria established by the American Society of Echocardiography (ASE) and the Society for Cardiovascular Angiography and Interventions (SCAI) (2015 edition), with right-to-left shunting (RLS) of grade II or higher upon Valsalva maneuver, as assessed by contrast-enhanced echocardiography;
5. Stable antiseizure medication regimen for at least four weeks prior to screening, with willingness to maintain a stable regimen throughout the study period;
6. At least one documented seizure episode during a six-week screening period (with a minimum of four weeks of effective seizure diary recordings) and a retrospective self-reported history of at least 12 seizures in the year preceding screening;
7. Ability to independently or with caregiver assistance complete a seizure diary and comply with clinical data collection and required medical examinations;
8. Willingness to undergo the investigational treatment and voluntary provision of written informed consent.

Exclusion Criteria:

1. Patients diagnosed with epilepsy of a known etiology, including infectious, metabolic, immune, genetic, or structural causes;
2. History of stroke or psychogenic nonepileptic seizures (PNES);
3. History of epilepsy surgery or implantable neurostimulation therapy, or planned epilepsy surgery, neurostimulation therapy, ketogenic diet therapy, or other antiseizure interventions during the study period;
4. Presence of structural cardiac abnormalities other than patent foramen ovale (PFO), such as moderate or severe valvular regurgitation or pulmonary hypertension;
5. Presence of severe central nervous system (CNS) diseases, including acute cerebrovascular disease, intracranial tumors, intracranial infections, or progressive CNS disorders;
6. Evidence of vascular puncture site infection or difficulty with puncture as assessed by transesophageal echocardiography combined with contrast-enhanced right heart echocardiography;
7. Documented contraindications to antiplatelet therapy;
8. Presence of severe psychiatric disorders, such as schizophrenia, bipolar disorder, or severe depression or anxiety;
9. History of alcohol or other substance abuse;
10. Severe dysfunction of vital organs (heart, lungs, liver, kidneys) deemed by the investigator to pose a risk to the participant or impair the participant's ability to complete the study;
11. Pregnant or breastfeeding women, or women planning to conceive during the study period;
12. Participation in another interventional clinical trial within three months prior to signing the informed consent form, current participation in another interventional trial, or plans to participate in another interventional trial during the study period; inability to comply with follow-up due to travel or relocation;
13. Any other condition that the investigator determines makes the patient unsuitable for participation in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage decrease in seizure frequency compared to baseline period | Week 48
  Percentage decrease in seizure frequency compared to baseline period

SECONDARY OUTCOMES:
Percentage decrease in mean duration of seizures from baseline period | Week 48
  Percentage decrease in mean duration of seizures from baseline period
Percentage of decrease from baseline in Epilepsy Severity | Week 48
  Percentage of decrease from baseline in Epilepsy Severity Scale score (NHS3)
Percentage improvement from baseline in Quality of Life for Patients with Epilepsy | Week 48
  Percentage improvement from baseline in Quality of Life Rating Scale for Patients with Epilepsy (QOLIE-31)
The maximum number of observation days without sustained epileptic seizures during the follow-up observation period | Up to 48 weeks
  The maximum number of observation days without sustained epileptic seizures during the follow-up observation period
The proportion of subjects whose seizure frequency decreased by more than 50% compared to the baseline period | Week 48
  The proportion of subjects whose seizure frequency decreased by more than 50% compared to the baseline period
The proportion of subjects whose average duration of epileptic seizures decreased by more than 50% compared to the baseline period | Week 48
  The proportion of subjects whose average duration of epileptic seizures decreased by more than 50% compared to the baseline period

OTHER OUTCOMES:
Scores of Hamilton Anxiety Scale (HAMA) | Week 24 and week 48
  The severity of anxiety
Scores of Hamilton Depression Scale (HAMD) | Week 24 and week 48
  The severity of depression
Scores of MMSE | Week 24 and week 48
  The severity of cognitive decline
Scores of MoCA | Week 24 and week 48
  The severity of cognitive decline
Scores of Headache Impact Test-6 | Week 24 and week 48
  The severity of migraine
Scores of Migraine-SpecificQuality-of-Life Questionnaire | Week 24 and week 48
  The severity of migraine
Scores of Pittsburgh Sleep Quality Index | Week 24 and week 48
  sleep quality
Incidence rate of adverse reactions | Up to 48 weeks
  Incidence rate of adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Westchina Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No